CLINICAL TRIAL: NCT05294497
Title: CSD201301: An In-Clinic Confinement Study to Assess Elements of Abuse Liability for Four P13 Nicotine Pouches
Brief Title: CSD201301: Study to Assess Elements of Abuse Liability for Four P13 Nicotine Pouches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CSD201301
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Smoking; Tobacco Use; Tobacco Smoking
MeSH Terms: conditions — Smoking; Tobacco Use; Tobacco Smoking | interventions — HTR3D protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Product usage order A B N C E D (Experimental): Subjects will use each of the 6 products sequentially (A B N C E D) during an evaluation period, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product N; Other: Product E
- Product usage order B C A D N E (Experimental): Subjects will use each of the 6 products sequentially (B C A D N E) during an evaluation period, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product N; Other: Product E
- Product usage order C D B E A N (Experimental): Subjects will use each of the 6 products sequentially (C D B E A N) during an evaluation period, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product N; Other: Product E
- Product usage order D E C N B A (Experimental): Subjects will use each of the 6 products sequentially (D E C N B A) during an evaluation period, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product N; Other: Product E
- Product usage order E N D A C B (Experimental): Subjects will use each of the 6 products sequentially (E N D A C B) during an evaluation period, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product N; Other: Product E
- Product usage order N A E B D C (Experimental): Subjects will use each of the 6 products sequentially (N A E B D C) during an evaluation period, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product N; Other: Product E

INTERVENTIONS:
Other: Product A — Usual Brand (UB) filtered, non-menthol or menthol cigarette
Other: Product B — Flavor variant P1312914 of a nicotine pouch product with 4 mg of nicotine
Other: Product C — Flavor variant P1312915 of a nicotine pouch product with 8 mg of nicotine
Other: Product D — Flavor variant P1313014 of a nicotine pouch product with 4 mg of nicotine
Other: Product N — Nicorette® White Ice Mint 4 mg nicotine gum
Other: Product E — Flavor variant P1313015 of a nicotine pouch product with 8 mg of nicotine

SUMMARY:
This is a two-site, open-label, randomized, 6-way cross-over study designed to evaluate elements of abuse liability (AL) including subjective effects and physiological measures (pharmacodynamics [PD]) and plasma nicotine uptake (pharmacokinetics [PK]) during and following ad libitum use of the study investigational products (IPs) by generally healthy smokers.

DETAILED DESCRIPTION:
Cigarette smokers and smokers also using smokeless tobacco products (ST) will be recruited into this AL study to evaluate elements of AL of four nicotine pouches compared to combustible cigarettes (CC) and nicotine polacrilex gum. At least one-third of the study population will include smokers using ST.

Potential subjects may complete a pre-screening telephone interview. They will complete a Screening Visit to assess their eligibility within 45 days prior to check-in and enrollment.

Starting on Day 1, subjects will check-in at the clinical site to complete procedures to confirm eligibility. Eligible subjects will be enrolled and confined for 7 days. Subjects will be randomized to one of 6 product sequences (using a Williams Design) in which they will evaluate one IP in each of six separate Test Sessions, such that each subject will evaluate six IPs, including four nicotine pouch IPs, and both a high-AL comparator (subject's usual brand [UB] cigarette) and a low-AL comparator (a commercially available nicotine replacement therapy [NRT] nicotine gum).

On Day 2 and continuing through Day 7, subjects will participate in Test Sessions that will last for approximately 4 hours. Each Test Session will include collection of both PD measures (subjective and physiological) and PK measures prior to, during and following IP use.

On the half day prior to each respective Test Session, a Product Acclimation Period will allow subjects ad libitum use of the randomized IP (at least two trial uses) for product familiarization prior to use in the next day's Test Session. Subjects can also use their UB cigarettes ad libitum, until the 12-hour tobacco abstinence begins prior to each Test Session, as long as the minimum use requirement for randomized IP is met.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an informed consent form (ICF) and complete questionnaires written in English.
2. Generally healthy males or females, 21 to 60 years of age, inclusive, at the time of consent.
3. Smokes combustible, filtered, non-menthol or menthol cigarettes, 83 mm to 100 mm in length as primary source of tobacco.
4. Smokes an average of at least 10 cigarettes per day (CPD) and inhales the smoke, for at least 6 months prior to Screening. Brief periods of abstinence due to illness, quit attempt (prior to 30 days of Screening), or clinical study participation (prior to 30 days of Screening) will be allowed at the discretion of the PI.
5. Smokers who also use ST products (e.g., moist snuff, snus), and have used ST within 30 days prior to screening will be enrolled.
6. Agrees to smoke the same UB cigarette throughout the study period. The UB cigarette is defined as the reported cigarette brand style currently smoked most frequently by the subject.
7. Expired breath carbon monoxide (ECO) level is ≥ 10 ppm and ≤ 100 ppm at Screening and at check-in Day 1.
8. Positive urine cotinine test at Screening.
9. Response at Screening to the Fagerström Test for Nicotine Dependence (FTND) Question 1 ("How soon after you wake up do you smoke your first cigarette?") is either "Within 5 minutes" or "6-30 minutes" (Heatherton et al., 1991).
10. Willing to use UB cigarette, nicotine pouch IPs, and Nicorette® gum during the study period.
11. Willing to abstain from tobacco and nicotine use for at least 12 hours prior to the start of each of six Test Sessions.
12. Females must be willing to use a form of contraception acceptable to the PI from the time of signing the informed consent until End-of-Study.

    Examples of acceptable means of birth control are, but not limited to:
    1. Surgical sterilization (hysterectomy, bilateral tubal ligation/occlusion, bilateral oophorectomy, bilateral salpingectomy);
    2. physical barrier method (e.g., condom, diaphragm/sponge/cervical cap) with spermicide;
    3. non-hormone releasing intrauterine devices (IUD) or hormone-releasing IUDs (e.g., Mirena or Kyleena);
    4. vasectomized partner; and
    5. post-menopausal and not on hormone replacement therapy.
13. Agrees to an in-clinic confinement of 7 days (6 nights).

Exclusion Criteria:

1. Presence of clinically significant uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, gastrointestinal, psychiatric, hematological, neurological disease, or any other concurrent disease or medical condition that, in the opinion of the PI, makes the study subject unsuitable to participate in this clinical study.
2. History, presence of, or clinical laboratory test results indicating diabetes.
3. Scheduled treatment for asthma currently or within the past consecutive 12 months prior to the Screening Visit. As-needed treatment, such as inhalers, may be included at the PI's discretion pending approval from the Medical Monitor.
4. History or presence of bleeding or clotting disorders.
5. Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that has been surgically and/or cryogenically removed.
6. Systolic blood pressure of > 160 mmHg or a diastolic blood pressure of > 95 mmHg, measured after being seated for five minutes at Screening and at check-in Day 1.
7. Weight of ≤ 110 pounds.
8. Hemoglobin level is < 12.5 g/dL for females or < 13.0 for males g/dL at Screening.
9. Females who have a positive pregnancy test, are pregnant, breastfeeding, or intend to become pregnant during the course of the study.
10. A positive urine drug screen without evidence of prescribed corresponding concomitant medication(s) at Screening or check-in Day 1.
11. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
12. Use of any medication or substance that aids in smoking cessation, including but not limited to any nicotine replacement therapy (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within (≤) 30 days prior to signing the informed consent.
13. Postpones a decision to quit using tobacco- or nicotine-containing products in order to participate in this study or self-reports a previous quit attempt within (≤) 30 days prior to signing the informed consent.
14. Any use of daily aspirin (≥ 325 mg) or any use of other anticoagulants.
15. Individuals ≥ 35 years of age currently using systemic, estrogen-containing contraception or hormone replacement therapy.
16. Whole blood donation within 8 weeks (≤ 56 days) prior to signing the informed consent and between Screening and check-in Day 1.
17. Plasma donation within (≤) 7 days prior to signing the informed consent and between Screening and check-in Day 1.
18. Employed by a tobacco or nicotine company, the study site, or handles tobacco- or nicotine-containing products as part of their job.
19. Participation in another clinical trial within (≤) 30 days prior to signing the informed consent. The 30-day window for each subject will be derived from the date of the last study event in the previous study to the time of signing the informed consent in the current study.
20. Drinks more than 21 servings of alcoholic beverages per week.
21. Has a positive alcohol result at Screening or check-in Day 1.
22. Determined by the PI to be inappropriate for this study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
(AUECPL) 5-240: area-under-the-effects curve (AUEC) for Product Liking (PL) | 5 minutes to 240 minutes
  area-under-the-effects curve (AUEC) for PL numeric rating scale (NRS) score-versus-time curve from 5 minutes to 240 minutes after the start of IP use. Product Liking is a numeric rating scale ranging from 0 to 10. A higher score indicates a higher liking of the product.
Emax PL: Maximum product liking (PL) | 240 minutes
  Maximum product liking (PL) numeric rating scale (NRS) score after the start of IP use. Product Liking is a numeric rating scale ranging from 0 to 10. A higher score indicates a higher liking of the product.

CONTACTS AND LOCATIONS:
Overall Officials: Milly Kanobe, PhD, Study Director — RAIS
Locations (2):
- United States (2):
  - AMR Lexington, Lexington, Kentucky
  - AMR Knoxville, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kanobe MN, Powell CY, Patrudu M, Baxter SA, Tapia MA, Darnell J, Prevette K, Gibson AG, Ayoku SA, Campbell L, Coffield JW, Keyser BM, Ganesh BS, Gale N, Jordan KG. Randomized crossover clinical studies to assess abuse liability and nicotine pharmacokinetics of Velo Oral Nicotine pouches. Front Pharmacol. 2025 Mar 13;16:1547073. doi: 10.3389/fphar.2025.1547073. eCollection 2025. PMID 40183092